CLINICAL TRIAL: NCT02365051
Title: Translation of COPE for Publicly-Funded Home Care Clients and Their Families
Acronym: COPECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Responsible Party: Principal Investigator, Fortinsky, Richard, Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-014-3
Record Dates: First submitted 2015-01-26; First posted 2015-02-18 (Estimated); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Dementia; Alzheimer's Disease
MeSH Terms: conditions — Dementia; Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- usual care (No Intervention): Older adults with dementia and their family caregivers receive all services for which they are eligible in the Connecticut Home Care Program for Elders.
- COPE plus usual care (Experimental): Older adults with dementia and their family caregivers receive Usual care plus the intervention: Care of Persons with Dementia in their Environments.
  Interventions: Behavioral: Care of Persons with Dementia in their Environments

INTERVENTIONS:
Behavioral: Care of Persons with Dementia in their Environments — In-home visits by occupational therapist and advanced practice nurse.
  Other Names: COPE
  Arms: COPE plus usual care

SUMMARY:
This community-based translational trial tests the value of a proven non-pharmacologic intervention for older adults living with dementia and informal caregivers when this intervention is incorporated into a publicly-funded home and community based service program. Half the participants will receive customary publicly-funded services alone, and half will receive customary services plus the proven non-pharmacologic intervention.

DETAILED DESCRIPTION:
More than 5 million Americans have dementia and more than 15 million Americans, mostly family members, provide unpaid care to these individuals. In the absence of a cure or widely effective pharmacotherapy to combat dementia, translation and implementation of efficacious non-pharmacologic interventions into existing service programs are sorely needed. The Connecticut Home Care Program for Elders (CHCPE), a Medicaid waiver and state revenue-funded program for older adults at high risk for nursing home admission, provides in-home and community-based services coordinated by care managers. In this translational study, an evidence-based intervention, Care of Persons with Dementia in their Environments (COPE), is incorporated into the CHCPE. COPE is an efficacious 4-month, in-home, non-pharmacologic intervention using occupational therapists and advanced practice nurses to maximize physical function in older adults with dementia and to improve dementia management skills of family caregivers (CG).

This trial will randomly assign 290 CHCPE clients with dementia and their CGs to receive either COPE plus customary CHCPE services, or customary CHCPE services alone. The main study outcome measures are similar to those of the original COPE efficacy trial. To maximize the translational effort, this study also will: conduct a formal cost-benefit analysis to determine the potential economic benefit of adding COPE to customary CHCPE services; evaluate the feasibility and acceptability of COPE as a new CHCPE service; and establish an expert Translational Advisory Committee to help develop and guide COPE dissemination plans for implementation nationally.

Study aims for CHCPE clients:

Aim 1.1: Determine COPE effect on functional dependence 4 months after randomization (primary study endpoint).

Aim 1.2: Determine COPE effects on engagement in activities, quality of life, and NPS, 4 months after randomization.

Aim 1.3: Determine COPE effects on functional dependence, engagement in activities, quality of life, and neuropsychiatric symptoms (NPS), 12 months after randomization.

We hypothesize that CHCPE clients receiving COPE will show greater reduction in functional dependence, greater engagement in activities, better quality of life, and fewer neuropsychiatric symptoms, compared to controls, 4 months and 12 months after randomization.

Study aims for CGs:

Aim 2.1: Determine COPE effect on perceived CG well-being 4 months after randomization.

Aim 2.2: Determine COPE effects on CG confidence in using dementia management strategies 4 months after randomization.

Aim 2.3: Determine COPE effects on CG perceived well-being, confidence in using activities, and ability to keep client at home, 12 months after randomization.

We hypothesize that COPE CGs will report improvement in all specified outcomes compared to controls, 4 and 12 months after randomization.

Translational study aims:

Aim 3.1: Determine the net financial benefit of COPE, accounting for COPE intervention costs, CHCPE usual care costs, nursing home costs, and other service costs, 4 months and 12 months after randomization. The 12 month cost-benefit analysis will test whether financial benefits of COPE accrue over a longer time horizon than the 4-month intervention period.

Aim 3.2: Determine the feasibility and acceptability of COPE implementation into the CHCPE from multiple stakeholder viewpoints, including CHCPE care managers and state Medicaid and public policy decision makers.

ELIGIBILITY:
Inclusion Criteria:

* Active client in publicly-funded home care program; Diagnosis of Alzheimer's disease or other dementia OR >=4 errors on the Mental Status Questionnaire; speaks or understands English

Exclusion Criteria:

* Diagnosed schizophrenia or bipolar disorder; bedbound; participation in experimental drug study to treat agitation; home environment deemed unsafe or unsanitary.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 582 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Functional dependence | Change in functional dependence score between baseline (pre-randomization) and 4 months post-randomization
  The metric for the primary outcome measure is score on the 15-item Caregiver Assessment of Function and Upset (CAFU) measure. The CAFU is adapted from the Functional Independence Measure; each of the 15 items is an activity of daily living (ADL) or instrumental activity of daily living (IADL). Each ADL and IADL item is scored on a 7-point scale ranging from completely independent (score of 7) to needing complete help (score of 1). Person-level functional dependence scores are calculated by summing scores across all items and dividing by the number of items.

CONTACTS AND LOCATIONS:
Overall Officials: Richard H Fortinsky, PhD, Principal Investigator — UConn Health
Locations (1):
- UConn Center on Aging, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Study results will be disseminated through peer-reviewed publications and presentations at national meetings in gerontology, geriatrics, public health, occupational therapy and nursing. Research-quality data which documents, supports and validates research findings will be made publicly available after main findings from the final research data set have been accepted for publication. Such data will be completely de-identified to prevent disclosure of individual study participant information, and will be shared on electronic media. We will request a data-sharing agreement that provides for a commitment to using the data only for research purposes, securing the data using appropriate computer technology, not redistributed to third parties, destroying or returning the data after analyses are completed, and a proper acknowledgement of the data resource.

REFERENCES:
- [Result] Fortinsky RH, Gitlin LN, Pizzi LT, Piersol CV, Grady J, Robison JT, Molony S. Translation of the Care of Persons with Dementia in their Environments (COPE) intervention in a publicly-funded home care context: Rationale and research design. Contemp Clin Trials. 2016 Jul;49:155-65. doi: 10.1016/j.cct.2016.07.006. Epub 2016 Jul 6. PMID 27394383
- [Result] Fortinsky RH, Gitlin LN, Pizzi LT, Piersol CV, Grady J, Robison JT, Molony S, Wakefield D. Effectiveness of the Care of Persons With Dementia in Their Environments Intervention When Embedded in a Publicly Funded Home- and Community-Based Service Program. Innov Aging. 2020 Oct 26;4(6):igaa053. doi: 10.1093/geroni/igaa053. eCollection 2020. PMID 33367114
- [Result] Pizzi LT, Jutkowitz E, Prioli KM, Lu EY, Babcock Z, McAbee-Sevick H, Wakefield DB, Robison J, Molony S, Piersol CV, Gitlin LN, Fortinsky RH. Cost-Benefit Analysis of the COPE Program for Persons Living With Dementia: Toward a Payment Model. Innov Aging. 2021 Oct 16;6(1):igab042. doi: 10.1093/geroni/igab042. eCollection 2022. PMID 35047708
- [Result] Kellett K, Robison J, McAbee-Sevick H, Gitlin LN, Verrier Piersol C, Fortinsky RH. Implementing the Care of Persons With Dementia in Their Environments (COPE) Intervention in Community-Based Programs: Acceptability and Perceived Benefit From Care Managers' and Interventionists' Perspectives. Gerontologist. 2023 Jan 24;63(1):28-39. doi: 10.1093/geront/gnac068. PMID 35581164